CLINICAL TRIAL: NCT06421922
Title: The Effects of Supplementation of Diet With Fiber or Probiotic Yogurt on the Intestinal Barrier Integrity in Individuals With Constipation-predominant Irritable Bowel Syndrome
Brief Title: Effect of Different Dietary Therapies on Intestinal Barrier Integrity in Patients With Irritable Bowel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gulhane Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Emine Nuket Unsal, PhD, Dietitian, Head of Clinical Nutrition Department, Gulhane Training and Research Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 50687469-799; 50687469-799 (Other Grant/Funding Number: TUEK)
Record Dates: First submitted 2024-05-08; First posted 2024-05-20 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Irritable Bowel Syndrome-IBS
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1-regular constipation diet (Active Comparator): Group 1 received a regular constipation diet (n=21)
  Interventions: Dietary Supplement: Group 1 received a regular constipation diet
- Group 2-soluble fiber (Active Comparator): group 2 received a constipation diet rich in soluble fiber (n=17)
  Interventions: Dietary Supplement: Group 2 received a constipation diet rich in soluble fiber
- Group 3-probiotic yogurt (Active Comparator): group 3 received a constipation diet with added probiotic yogurt (n=22).
  Interventions: Dietary Supplement: Group 3 received a constipation diet supplemented with probiotic yogurt.

INTERVENTIONS:
Dietary Supplement: Group 1 received a regular constipation diet — Group 1 received only regular constipation diet, the constipation diet included 2 litres of water, 2 portions of vegetables, 3 portions of fruits and legumes 2 times a week. Followed 8 weeks.
  Arms: Group 1-regular constipation diet
Dietary Supplement: Group 2 received a constipation diet rich in soluble fiber — Soluble fiber (resistant starch) (5 g/day) was added to the constipation diet in group 2 as 1 sachet/day (5 g/day) during the initial 4 weeks and 2 sachets/day (10 g/day) in the following 4 weeks.
  Arms: Group 2-soluble fiber
Dietary Supplement: Group 3 received a constipation diet supplemented with probiotic yogurt. — "Bifidobacterium İnfantis 35624 (B. İnfantis 35624)" strain, which is specific to IBS, was added to yogurt in group 3, consumed before the lunch. The follow-up period was 8 weeks.
  Arms: Group 3-probiotic yogurt

SUMMARY:
This study aims to evaluate the effects of different dietary treatments on intestinal integrity in female subjects aged 19-50 years previously diagnosed with constipation-predominant irritable bowel syndrome (IBS). At the Gülhane Training and Research Hospital's gastroenterology clinic in Ankara, Turkey, a randomized controlled experiment was carried out. 60 individuals with IBS were randomly divided into three groups. Group 1 was assigned to a regular constipation diet, group 2 to a constipation diet rich in soluble fibers, and group 3 to a constipation diet with probiotic yogurt supplementation. Every individual was monitored for eight weeks. Plasma zonulin level was used to measure intestinal integrity both before and after treatment.

DETAILED DESCRIPTION:
This was a non-pharmacological randomized controlled trial conducted at Ankara Gülhane Training and Research Hospital Gastroenterology Polyclinic between June 2019 and March 2020. Participants of this study were women aged 19 to 50 years with a diagnosis of IBS according to the Rome IV criteria (2017).

The sample size was calculated with G*Power software. With an estimated power of 90%, a Type I error of 0.05, and an effect size of f=0.25, the total sample size required was 54, consisting of 18 participants in each group. The sample size was calculated using G*Power software. The total sample size, with an estimated strength of 90%, Type I error of 0.05, and effect size f = 0.25, was 54, consisting of 18 participants in each group. 60 participants were targeted due to compensation for potential drop-out from protocol.

Using random assignment software, participants were divided into three groups at random for parallel group randomized trials. Group 1 received a standard constipation diet; Group 2 received a soluble fiber-rich constipation diet; and Group 3 received a probiotic yogurt-supplemented constipation diet. The three groups-regular constipation diet, constipation diet high in soluble fiber, and constipation diet fortified with probiotic yogurt-were coded R 1-2, F 1-2, and P 1-2 to protect patient confidentiality. Twice a week, two liters of water, two servings of vegetables, and three servings of fruits, and legumes were the staples of the constipation diet. For the first four weeks, Group 2's constipation diet included 1 sachet of soluble fiber (resistant starch) (5 g/day), and in the second week, 2 sachets of soluble fiber (10 g/day) were added. It happens after four weeks. In Group 3, the yogurt ingested before lunch was supplemented with the IBS-specific strain "Bifidobacterium Infantis 35624 (B. Infantis 35624)". For eight weeks, there was a follow-up.

All data were collected by face-to-face survey method. At the first visit, sociodemographic characteristics and three-day food consumption were recorded. Food consumption was recorded for 3 days, 2 days on weekdays, and 1 day on weekends. Serum Zonulin level and biochemical tests were evaluated at the beginning of the diet and the 8th week. Serum Zonulin level was measured using the "BT Lab Human Zonulin ELISA Kit" (China, E1117). Daily energy and nutrient amounts taken from the diet were analyzed using the Nutrition Information System 8 (BeBis 8) computer package program.

IBM SPSS Statistics 22.00 program was used to analyze the data obtained. The normal distribution of the data was evaluated with the Shapiro-Wilk test. To increase clarity and ensure consistency with other studies, continuous variables are presented as mean ± standard deviation. Spearman rank correlation coefficients are a way to represent correlations between continuous variables. Analysis of variance or the Kruskal Wallis test was used to compare groups. Wilcoxon signed-rank test was used to compare groups within the same group from baseline to week eight. The significance threshold of p<0.05 was determined.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 19-50 years who were diagnosed with IBS according to Rome IV criteria
* Any metabolic disease (diabetes, heart disease, etc.), cancer and autoimmune no history of chronic diseases such as illness
* Not being pregnant or lactating
* Body mass index (BMI) of 18.5-29.9 kg/m2

Exclusion Criteria:

* Chronic disease history such as cancer and autoimmune diseases
* Probiotics use or nutritional supplement use (vitamins, minerals) in the last 6 months.
* Pregnancy.

Ages: 19 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 60 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2019-10-15 (Actual); Study Completion 2020-06-07 (Actual)

PRIMARY OUTCOMES:
Serum Zonulin level | 0-8 weeks
  The primary outcome was the change in blood Zonulin level after adding probiotic yogurt to a regular constipation diet instead of soluble fiber. Serum zonulin levels were analysed to evaluate the effect of dietary compliance on intestinal barrier integrity. Lower serum zonulin levels indicate a better intestinal barrier integrity.

SECONDARY OUTCOMES:
Other biomarkers (fasting blood glucose, cholesterol, blood triglyceride, LDL cholesterol and CRP) | 0-8 weeks
  The secondary outcomes were changes in fasting blood glucose, cholesterol, blood triglyceride, LDL cholesterol and CRP levels after adding probiotic yogurt to a regular constipation diet instead of soluble fiber.

CONTACTS AND LOCATIONS:
Overall Officials: Emine Nuket Unsal, Phd, Principal Investigator — Gulhane Training and Research Hospital
Locations (1):
- GulhaneTRH, Ankara, Keçiören, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No